CLINICAL TRIAL: NCT03994172
Title: Novel Combination Therapy for Osteoporosis in Men
Acronym: Osteo-Men
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDB-012-17F; 1 IO1 CX001514-01A2 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Male Osteoporosis
Keywords: male osteoporosis; anabolic therapy; teriparatide; calcimimetic; calcium-sensing receptor; PTH receptor; bone formation
MeSH Terms: interventions — Teriparatide; PTH protein, human; Cinacalcet; Calcium Citrate; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: The study design is that of a randomized double-blind, placebo (PBO)-controlled trial of the combination of teriparatide (TPTD) + the calcimimetic cinacalcet compared to monotherapy with TPTD alone in men with low bone mineral density (BMD).
Who Masked: Participant, Care Provider, Investigator
Masking Description: All study personnel will be masked to treatment assignment and this group will include the DXA technicians, the study coordinators, and the lab technicians and lab supervisors who will analyze samples for study results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- teriparatide (TPTD) + the calcimimetic cinacalcet (Experimental): Combination arm: Men randomized to this arm will take daily subcutaneous injections of teriparatide [PTH (1-34)] (20 mcg per day) and at the same time swallow a 30-mg tablet of cinacalcet. Men in both arms of the study will take a total of approximately 1000 mg elemental Ca through their diets and study provided Ca supplements (Ca citrate) and approximately 1000 IU vitamin D3. Men will be followed and assessed throughout the entire study using the clinical (vital signs, adverse events), laboratory (blood and urine tests) and densitometric procedures (DXA BMD and TBS) outlined in the study protocol.
  Interventions: Drug: Teriparatide or human parathyroid hormone (PTH) 1-34; Drug: Cinacalcet; Dietary Supplement: Calcium citrate tablet; Dietary Supplement: Vitamin D3
- teriparatide (TPTD) + placebo (Placebo Comparator): Monotherapy arm: Men randomized to this arm will take daily subcutaneous injections of teriparatide [PTH (1-34)] (20 mcg per day) and at the same time swallow a placebo tablet. Men in both arms of the study will take a total of approximately 1000 mg elemental Ca through their diets and study provided Ca supplements (Ca citrate) and approximately 1000 IU vitamin D3. Men will be followed and assessed throughout the entire study using the clinical (vital signs, adverse events), laboratory (blood and urine tests) and densitometric procedures (DXA BMD and TBS) outlined in the study protocol.
  Interventions: Drug: Teriparatide or human parathyroid hormone (PTH) 1-34; Drug: placebo tablet; Dietary Supplement: Calcium citrate tablet; Dietary Supplement: Vitamin D3

INTERVENTIONS:
Drug: Teriparatide or human parathyroid hormone (PTH) 1-34 — Teriparatide or PTH 1-34 is a 34 amino acid peptide derived by recombinant DNA technology from the authentic sequence of human parathyroid hormone. It is given by subcutaneous injection in the dosage of 20 micrograms per day in the trial in both treatment arms for the 48 weeks or 11 months of the trial.
  Other Names: Forteo
Drug: Cinacalcet — This drug is an orally active calcimimetic (drug that activates Ca-sensing receptors on target cells) that will be given daily orally to the men randomized to the Experimental Treatment Arm (#1). Cinacalcet tablets will be given simultaneously with the injection of PTH(1-34) or teriparatide. Cinacalcet will be given only once daily but given every single day of the trial starting with the Randomization Visit for the duration of 48 weeks or 11 months of the trial.
  Other Names: Sensipar
  Arms: teriparatide (TPTD) + the calcimimetic cinacalcet
Drug: placebo tablet — The placebo tablet in the trial will be purchased from Consolidated Midland Corporation in Brewster, NY. Each white tablet contains Lactose, Stearic Acid and Magnesium Stearate (330 mg total). Subjects randomized to the placebo arm or Placebo - Arm #2 - will take one tablet orally at the same time as he injects the teriparatide each day. Placebo tablets will be given only once daily but given every single day of the trial starting with the Randomization Visit for the duration of 48 weeks or 11 months of the trial.
  Other Names: placebo
  Arms: teriparatide (TPTD) + placebo
Dietary Supplement: Calcium citrate tablet — Ca citrate supplements (forms 200 or 250 mg elemental Ca/oral tablet) will be used in the study. Each subject will have average dietary Ca intake quantified by a Food Frequency Questionaire. Each subject will take sufficient Ca citrate supplements to make the total Ca intake equal ~1000 mg per day (diet+supplements). Ca supplements will be spread out during the day so that any amount of supplements over 500 mg will be taken at 2 different time-points. Ca citrate supplements will be sourced by our research pharmacist will be of high-quality and consistency. Ca supplements will be started at Screening Visit 2 and given for a 4-week run-in period. Once subjects are randomized to Arm 1 or Arm 2 of the trial, subjects will continue to take daily Ca supplements at the same dose and times as during the run-in period. That daily dosing will continue from day of Randomization through the end of 48 weeks or 11 months of the trial.
  Other Names: Calcium citrate supplement
Dietary Supplement: Vitamin D3 — Subjects will be given 1000 IU vitamin D3 in tablet form to be taken orally once a day at any time during the day. Vitamin D3 supplements will be sourced by our research pharmacist and supplements selected for use in the trial will be of high quality and consistency. Vitamin D3 supplements will be started at Screening Visit 2 in the trial and given for a 4-week run-in period. Once subjects are randomized to Arm 1 or Arm 2 of the trial, subjects will continue to take daily vitamin D3 supplements at the same dose and timing as during the run-in period. That daily dosing will continue from the day of Randomization Visit through to the end of the 48 weeks or 11 months of the trial.
  Other Names: Cholecalciferol

SUMMARY:
Osteoporotic fractures are a key health problem in older men. Although there are drugs approved to treat osteoporosis in men [bisphosphonates, denosumab, and teriparatide (TPTD) or PTH(1-34)], there is a lack of knowledge on how to use them effectively. TPTD is a potent bone anabolic drug, meaning that it builds bone mass. However, doctors do not know if it should only be used as single drug or whether it can be more effectively combined to achieve the most benefit? This trial will test a novel combination therapy for osteoporosis in men based on exciting laboratory findings in mice. TPTD works to raise bone mass and improve bone strength by stimulating PTH receptors (PTH-Rs) on the membranes of bone-forming cells or osteoblasts (OBs). Calcimimetics are drugs that activate calcium receptors (CaSRs) in OBs. CaSRs in OBs participate in new bone formation. Daily injections of TPTD, given along with a calcimimetic drug (called NPS-R568), over 6 weeks markedly improved bone mineral density (BMD) and structure in mice. This study will test whether the combined activation of PTH-Rs and CaSRs (by the combination treatment of TPTD+calcimimetic cinacalcet) in men will produce greater bone forming responses than PTH-R activation alone (TPTD+placebo). The study has two aims and will be done in 48 men with low bone mass: (1) to determine the effects of 11 months treatment with TPTD+cinacalcet vs TPTD+placebo on BMD and bone metabolism by assessing lumbar spine BMD (primary endpoint), femoral neck BMD, and levels of the bone formation marker serum N-terminal pro-peptide of type 1 collagen; (2) to determine the biochemical responses by blood tests in men who receive the combination of TPTD+cinacalcet compared to men who get TPTD+placebo treatment. This is done by quantifying acute and chronic changes in serum calcium and PTH levels right after these drugs are given and how much calcium is excreted in the urine over time, with both treatment regimens. This study will help to understand whether an effective combination therapy in mice will prove to be effective in men.

DETAILED DESCRIPTION:
NOVEL COMBINATION THERAPY FOR OSTEOPOROSIS IN MEN

1. Background for the Study

   What Is the Risk of Osteoporotic Fractures in Men and Why Do Men Lose Bone Mass? Osteoporosis is a neglected condition in men. Yet, men sustain approximately 30% of the 1.5 million fractures that occur annually in the US. Fractures are expensive. Estimated costs are at least $20 billion annually. This figure will no doubt rise substantially as the population ages. Plus, these costs do not take into account the personal and societal burden of fractures, especially hip fractures. One in 6 men will sustain a hip fracture by the time he reaches age 90 years. A man who fractures a hip at any age has greater disability following that fracture and is much less likely to regain his ability to walk and to live independently afterward. Men also have a greater risk of dying from the complications of hip fractures. Overall, one-year mortality for patients who sustain a hip fracture is ~20%. However, mortality in men with hip fractures is staggeringly high at ~37.5% in the first year.

   The pathophysiology of bone loss in aging men differs in important ways from postmenopausal osteoporosis. Age-related bone loss in men begins in the 6th decade with nutritional and hormonal abnormalities playing important roles. Contributing factors include decreased intestinal Ca absorption, vitamin D deficiency or insufficiency, and secondary (2o) hyperparathyroidism (HPT). Testosterone levels decline with age in men, and as they do, estradiol levels also fall. Considerable evidence supports an important role for estradiol in maintaining bone mass in men as well as women. Men lose both trabecular and cortical bone mass with age. Trabecular bone thins out in men, rather than perforates, as it does in women, and excessive cortical bone remodeling is a dominant force in older men. In men, periosteal bone apposition does not keep pace with endosteal resorption, and the bones weaken. With minimal trauma, fragility fractures may result. Thus, reduced bone formation is a key mechanism underlying bone loss in men, more so than the high rates of bone resorption seen in postmenopausal estrogen deficiency. For these reasons, anabolic regimens that enhance bone formation may achieve better clinical outcomes in men compared to commonly used antiresorptive agents. This trial will test a novel anabolic combination therapy in men.

   How Effective Are Current Treatments for Osteoporosis in Men? Several agents have been Food and Drug Administration (FDA)-approved to treat osteoporosis in men: bisphosphonates; denosumab; and teriparatide (TPTD) or parathyroid hormone (PTH) (1-34). In trials enrolling men, these agents were shown to increase bone mineral density (BMD) by dual energy Xray absorptiometry (DXA) at key skeletal sites, quantitatively similar to their effects in postmenopausal women. In only a few appropriately powered studies, there was a reduction in incident vertebral fractures in men at high risk and/or those on androgen deprivation therapy.

   Intermittent injections of TPTD are appealing as a treatment for osteoporosis in men because the agent has potent anabolic actions. TPTD increases bone formation, reflected by enhanced biochemical markers of osteoblast (OB) activity, such as N-terminal propeptide of type 1 collagen (P1NP) and bone specific alkaline phosphatase (BSAP) in the blood, and by direct histomorphometric quantification of bone formation, and mineral apposition rates. TPTD also improves the microarchitecture of bone by micro-CT (trabecular thickness and connectivity) and increases the maturation or number of circulating osteogenic precursors and stem cells in blood in postmenopausal women. TPTD in vitro stimulates the proliferation of mesenchymal stem cells and their commitment to the OB lineage as osteoprogenitors. PTH (1-34) also increases differentiation of early OBs and matrix production, blocks apoptosis of OBs and osteocytes, and reduces production of the Wnt inhibitor sclerostin by osteocytes. The anabolic actions of PTH treatment within a defined time-frame (18 to 24 months in humans) -- called the "anabolic window" -- improve bone strength and ultimately reduce spine and nonvertebral fractures. Over time, however, PTH stimulates receptor activator of nuclear factor kappa B ligand (RANK-L) production by early OB lineage cells, and RANK-L enhances osteoclast (OC) production. This increases bone resorption, which limits further gains in BMD with PTH. The challenge in designing optimal treatment regimens with PTH is maximizing its anabolic activity, while taming its catabolic effects on bone.

   Clinical trials with TPTD [recombinant human PTH (1-34)] or synthetic human PTH (1-34) in men are limited to a few studies with small numbers of men. Orwoll and colleagues randomized 437 men into 3 groups: placebo (PBO) vs 20 (the dose subsequently FDA-approved) or 40 ug TPTD daily. However, they completed only an average of 11 months on treatment. Kurland and colleagues randomized 23 men to synthetic PTH (1-34) (400 IU or ~25 ug/day; N=10) or PBO (N=13) for 18 months. Finkelstein and colleagues, as part of a combination study, randomized 27 men to synthetic PTH (1-34) for 24 months (37 ug/day). Thus, that study used twice the approved dose of PTH (1-34). Walker and colleagues randomized men to risedronate (35 mg/week) (N=10), TPTD (20 ug/day) (N=9), or the combination (N=10) for 18 months. In these studies, BMD rose by ~6-14% at the lumbar spine and by ~2-4% at femoral neck with 11-18 months treatment [with 20 or 25 ug PTH (1-34)/day]. Higher doses of PTH (1-34) (37 or 40 ug/day) produced even greater responses at both sites (2-3 fold more). This indicates that stronger anabolic effects are feasible to achieve in men within these short time-frames. However, these doses are less tolerated, and the investigators do not plan to use them. Rather, the trial proposed will use the FDA-approved dose of TPTD (20 ug/d) by daily subcutaneous injection.

   Combination studies of PTH (1-34) with alendronate or TPTD with risedronate did not convincingly show synergistic effects on BMD in men. A trial combining TPTD and denosumab showed additive effects of the combination, but it was done in women. Several important questions about TPTD treatment in men have never been addressed. Among them, can TPTD be advantageously combined with another "bone-active" drug that has a similar or a different mechanism of action? Investigators in the field only know that adding PTH (1-34) to alendronate in men does not produce additive effects. This trial will test the hypothesis that concurrent CaSR activation (by calcimimetic) synergizes with PTH-R activation (by TPTD) to produce greater anabolic effects in men, reflected by changes in BMD and bone turnover markers (BTMs), compared to TPTD alone. This is a novel combination therapy that is well-supported in preclinical studies.
2. Scientific Premise for the Planned Intervention This is a first in human study of a combination therapy for osteoporosis. Both of the drugs that will be used in the trial have been FDA-approved for many years and have been used in the clinic in hundreds of thousands of patients worldwide: TPTD for the treatment of osteoporosis in women and men, and cinacalcet for the treatment of various forms of HPT in women and men. The two agents to be used in the trial have not been as yet tested in the combination format that will be done in this study.

   Summarized below are preclinical data from young (12-week old) and elderly (12-month old) male and female mice.

   Preclinical Studies: Combined PTH(1-34) and Calcimimetic Produce Marked Anabolic Effects on Bone in Mice Both extracellular Ca-sensing receptors (CaSRs) and PTH receptors (PTH-Rs) play central roles in the control of bone remodeling. In conditional (or tissue-specific) knockout mice, CaSRs have been shown to play key roles in skeletal development and in OB and osteocyte function by several groups. Such work supports the idea that high extracellular [Ca] ([Ca]e), acting through CaSRs, is an "anabolic pathway" in bone, akin to intermittent PTH (1-34) stimulation of PTH-R signaling in bone. Several groups have found that direct CaSR activation in OC lineage cells reduced their survival, gene expression, and resorptive function. This suggested that enhanced OB and suppressed OC function might be accomplished through activation of CaSRs in different bone cell populations.

   Based on this work in mice and the known role of PTH peptides as bone anabolic agents in humans, studies were done in mice to test the hypothesis that concurrent activation of PTH-Rs and of CaSRs has synergistic effects on bone mass. Adult male mice given intermittent subcutaneous (SC) injections of PTH(1-34) (40-80 ug/kg) and the calcimimetic NPS-R568 (20 umole/kg) for 4-6 weeks showed dramatic synergistic anabolic effects on bone mass and strength. PTH (1-34) injections alone significantly increased trabecular (Tb) bone mass [Tb bone volume/tissue volume (BV/TV)] by micro-CT in the distal femur as well as Tb thickness (TbTh) (p<0.05). Co-injections of PTH (1-34) and NPS-R568 produced significantly greater effects on Tb BV/TV and TbTh (by ~21%; p<0.01), while NPS-R568 injections alone had no effect. These are large effects on bone mass, as determined by highly sensitive methods - micro CT and bone histomorphometry. The latter is the gold-standard for testing the effects of an intervention on dynamic bone metabolic processes. This combination therapy also produced bone microarchitectural changes (more plate-like trabeculi), compatible with mechanically stronger bone.

   Cortical (Ct) bone is typically less affected by PTH (1-34) treatment. However, in these experiments when Ct bone at the tibiofibular junction (TFJ) was assessed by micro-CT, it was clear that combined injections of PTH (1-34) and NPS-R568 produced dramatic increases in CtTV, CtBV, and CtTh of 8-10% (p<0.05). Thus, this work demonstrated clear "anabolic synergy" of concomitant PTH-R and CaSR activation on both Tb and Ct bone in adult male mice - findings potentially clinically significant and highly relevant to the proposed trial. Similar and dose-dependent increases were seen in Tb bone of the L5 vertebrae [in BV/TV, TbTh, and Tb number (N); p<0.05 or p<0.01] and in their Ct bone at the TFJ (CtTV, CtBV, and CtTh; p<0.05) in elderly female mice.

   Dynamic histomorphometry on bone biopsy specimens in the mice supported these results. Daily injections for 6 weeks of TPTD alone induced substantial bone formation by fluorescent tetracycline labelling from Ct bone sections. Bone formation was substantially augmented by co-administration of calcimimetic NPS R568. Quantitative analyses of Tb and Ct bone parameters (N=12 mice/group) supported the micro-CT data, indicating robustly strong increases in bone mass with this combination. By mechanical testing of the mouse femurs, bone strength was tested, and the bones were found to be stronger (greater energy to failure) in the male mice treated with combined PTH/NPS-R568 vs PTH (1-34)+vehicle.
3. Study Rationale Osteoporosis and fracture-related disability are important health problems in older men. Fractures increase mortality. Men who fracture their hips have twice the mortality of women sustaining those same hip fractures. Several drugs are approved to treat osteoporosis in men [bisphosphonates, denosumab, and teriparatide (TPTD) or PTH(1-34)], but there have been little insight as to how to use them most effectively. TPTD has great appeal for treating osteoporosis in men because it substantially improves bone mass, rebuilds the microarchitecture, improves bone strength, and reduces fractures. Little is known about the best ways to employ TPTD in the treatment of male osteoporosis. Should it be used only as monotherapy or does concurrent or sequential use with other agents lead to the greatest benefit? The proposed clinical trial is an effort to test a novel combination therapy for osteoporosis in men based on exciting preclinical findings in mice. It is known that TPTD achieves its anabolic effects by stimulating PTH-Rs in cells of the OB lineage. Calcimimetics mimic the effects of high extracellular calcium concentrations ([Ca]e) by activating CaSRs expressed in many cell types including OBs and OCs in bone.

   A.Specific Aims and Hypotheses Tested To address the hypothesis that concurrent CaSR and PTH-R activation produces synergistic anabolic effects on bone, a double-blind, PBO-controlled trial in 48 men with low BMD testing a novel combination regimen will be performed. Older male Veterans with low BMD by DXA will be randomized to 2 treatment arms: TPTD+cinacalcet vs TPTD+PBO. Efficacy endpoints will be changes in BMD by DXA and the bone turnover marker (BTM) P1NP (Aim 1). Pharmacodynamic (PD) effects of the combination regimen vs monotherapy will be profiled (serum Ca, PTH) and safety confirmed (Aim 2). A subset of 24 patients (12/treatment arm) will undergo detailed acute (8 hr) PD assessments and clinical monitoring at the UCSF CRC (Clinical Research Center). Safety will be assessed in all trial subjects with serum Ca and 24-hour urinary Ca monitoring and with adverse event (AE) and clinical assessments. Although both drugs used in this trial are FDA-approved (TPTD, 20 ug/day for osteoporosis; cinacalcet, 30 mg/day for HPT), an IND (Investigational New Drug) application is in place to give this drug combination.

   B.Study Aims and Hypotheses AIM 1: To determine the effects of treatment with TPTD+cinacalcet compared to TPTD+PBO on BMD and bone metabolism in men with low bone mass by assessing responses in lumbar spine (LS) BMD (primary endpoint) and femoral neck (FN) BMD and levels of P1NP.

   There are 2 hypotheses tested in this aim. Hypothesis 1a proposes that BMD responses to combined TPTD+cinacalcet are greater than those induced by TPTD+PBO. LS BMD typically responds quickly and robustly to TPTD and is the 1o endpoint of the trial. Changes in FN BMD, a site often slower to respond and with smaller magnitude, are a 2o endpoint. DXA measurements will be performed and analyzed as described below. Subjects will be treated for 11 months (48 weeks). All subjects will receive Ca and vitamin D3 supplements throughout the trial. Hypothesis 1b proposes that bone formation marker P1NP increases to a greater extent with combined TPTD+cinacalcet vs TPTD+PBO. P1NP is the best validated biomarker of TPTD action and responds rapidly and robustly to anabolic therapy, the change in P1NP at 3 months (12 weeks) after initiation of treatment is a key 2o endpoint for the study.

   AIM 2: To determine the pharmacodynamic (PD) responses to study drug administration in men with low bone mass by assessing acute and chronic changes in the serum [Ca] and plasma intact PTH after drug administration and changes in urinary Ca excretion.

   There are 2 hypotheses tested in the PD studies in this aim, which is focused on establishing physiologic responses and confirming safety with this combination therapy. Hypothesis 2a proposes that the serum [Ca] does not fall to >5% below the lower limits of the normal range in response to the administration of study drugs. After randomization, subjects will initiate dosing with the 2 study drugs. First, baseline sampling (pre-study drug) will be done, and then subjects will have blood collected for serum [Ca], albumin, and PTH at specific time-points in the 8 hours after study drugs are administered. As is clear from the literature on PTH actions in vivo, TPTD tends to raise serum [Ca], while cinacalcet is expected to lower intact PTH and thereby serum [Ca] usually transiently. It is anticipated that the effects of these 2 drugs, known to act over similar time-courses in humans, will tend to offset each other, so that the serum [Ca] remains stable and within the normal range in subjects taking the combination (TPTD+cinacalcet). In general, the majority of patients taking TPTD and the majority of those receiving cinacalcet should experience offset of drug effects well before 24 hours have elapsed post-dosing. Based on these kinetics, it is not expected that combined treatment will produce major steady-state changes in serum [Ca]. At the very least, it is expected that any serum [Ca] lowering will be modest (and transient), and steady-state levels will not drop >5% below the lower limit of the normal range. This will be carefully assessed, both acutely in the PD study [in 24 subjects (12/treatment arm)] and chronically by examining pre-dose serum [Ca] over the full study (in all subjects). Intact PTH will be monitored as an exploratory endpoint, since serum PTH levels may fall with chronic cinacalcet treatment. Determining changes in endogenous PTH secretion may be important for fully understanding the PD of concurrent TPTD+cinacalcet therapy.

   Hypothesis 2b proposes that urinary Ca excretion does not exceed 350 mg/24 hours in subjects receiving study drugs. This parameter will be carefully studied throughout the trial for these reasons. First, TPTD may raise urinary Ca because of increased gut Ca absorption [due to increased 1,25(OH)2 vitamin D] and enhanced Ca mobilization from bone (direct PTH action). Both effects increase the filtered load of Ca, which can raise urinary Ca. Second, calcimimetics, by stimulating renal CaSRs may also raise urinary Ca levels. Hypothesis 2b is predicated on the observation that men treated with TPTD alone did not excrete >350 mg Ca/24 hours according to prior clinical trial data. In addition, prior studies in patients with 1o HPT did not show significant hypercalciuria due to cinacalcet. However, data on urinary Ca in normal subjects taking calcimimetics are scant. If chronic hypercalciuria results from the combination therapy, there is potential for consequences (renal stones, possibly renal insufficiency) that will be key to know about. Thus, urinary Ca assessments throughout the study are critical safety endpoints.

   C.Primary and Secondary Objectives As primary objective, the study will examine the effects on LS BMD by DXA of treatment with the combination of TPTD (PTH 1-34) + placebo vs TPTD + oral calcimimetic cinacalcet in men with low bone mass or osteoporosis.

   The study has two secondary objectives: (1) assess the effects of combination of TPTD (PTH 1-34) + placebo vs TPTD + oral calcimimetic cinacalcet on FN BMD by DXA in men with low bone mass or osteoporosis; and (2) assess the effects of the combination of TPTD (PTH 1-34) + PBO vs TPTD + oral calcimimetic cinacalcet on the bone formation marker serum P1NP in men with low bone mass or osteoporosis.

   A safety assessment will include determining (a) acute and chronic changes in the concentrations of serum Ca ([Ca]) and plasma intact PTH after administration of study medications in both treatment arms in an 8 hour PD study; and (b) changes in 24 hour urinary Ca excretion (over full 11 month trial) with both treatment regimens.
4. Study Design and Protocol

A.Subjects There will be 48 men randomized to one of two treatment arms: TPTD + PBO tablet (N=24) or TPTD + cinacalcet tablet (N=24). Men of all ethnic and racial groups will be encouraged to participate. The DXA scan done at screening will be used to determine whether or not a man meets BMD criteria for enrollment into the study.

B.Inclusion and Exclusion Criteria for Subjects - described elsewhere in the application

C.Study Drugs and Supplements Teriparatide (TPTD) or PTH 1-34 which will be obtained from commercial sources and given at 20 mcg daily, by SC injection. Cinacalcet or sensipar, an oral calcimimetic, will be given at the dose 30 mg daily orally.

The PBO control will be a purchased "placebo" tablet that will be packaged in exactly the same manner as cinacalcet. Supplements in the form of Ca citrate tablets (200 or 500 mg tablets) will be given in both treatment arms to subjects along with vitamin D3 (1,000 International Units) by mouth daily. Ca supplements will be adjusted along with an assessment of dietary Ca intake to reach a total of ~1,000 mg elemental Ca per day.

D.Study Measurements Several types of measurements will be made in the course of the trial.

1. BMD will be measured at the LS, hip and radius by DXA at the UCSF CTSI CRC. Trabecular bone score (TBS) will also be determined from the data collected during the DXA assessment of the lumbar spine using commercially available software applications available at the investigators' center.
2. Biochemical markers of bone turnover (BTMs) and vitamin D metabolites will be measured during the study visits including the following: serum P1NP, serum C-telopeptide (CTX), bone specific alkaline phosphatase (BSAP), osteoprotegerin (OPG), RANK-L, and 1,25 (OH)2 vitamin D.
3. Dietary Ca intake will be assessed by the Block Food Frequency Questionnaire.
4. There will be PD testing during the study. This will include assessing acute changes in the serum levels of Ca, albumin, phosphate and PTH during the acute administration of the study drugs during an 8-hour PD test in the clinic at the Randomization Visit of the study; determining chronic changes in the serum levels of calcium and PTH during the entire study with the administration of the study drug combinations (11 months of the trial); studying chronic changes in the urinary calcium at study visits during the full trial.
5. In exploratory studies, peripheral blood mononuclear cells (PBMCs) will be collected by blood sampling of participants and those samples fractionated for cells of the OB and OC lineage to determine whether the two treatment interventions alter the levels and properties (gene expression markers) of the circulating populations of these cells.

   E.Study Duration and Study Visits Subjects will be on study for approximately 12-13 months. Screening will be conducted at 2 separate visits. This will be followed by a run-in period of 4 weeks for eligible subjects. The intervention period will be 11 months (48 weeks) in duration.

   Screening will be done through a telephone call to initiate contact, describe the study, and set up a visit to achieve informed consent and to do the screening DXA scan. There are two Screening Visits, the first will involve obtaining the DXA scan, and the second will involve lab testing, a complete medical history and physical exam to be performed. The run-in period during which the participant takes only calcium and vitamin D supplements for 4 weeks will follow.

   The Randomization Visit will involve lab testing and in 12/24 subjects in each arm, an 8-hour PD Study. Subjects will be randomized to one of the study treatment arms and taught to take the daily injections and the study medication tablets (cinacalcet vs PBO) At week 1, subjects will have lab testing done and a telephone visit. Thereafter, at Weeks 4, 8, 12, 20, 24, 36, and 48 there will be lab testing of blood and urine, assessment of adverse events, and clinical followup done. At the final visit (Week 48, approximately 11 months), a followup DXA scan will be done.

   F.Timeline of main study procedures and interventions (Mo=month)

   Screening Visit 1

   -Informed consent, DXA/TBS

   Screening Visit 2

   -History, physical exam, vital signs, screening labs (blood, urine), food frequency questionnaire, AE, concomitant medications, pen teaching, supplements dispensed

   Randomization Visit -PD study, vital signs, labs (blood, urine), AE, concomitant medications, pen teaching, supplements and study drugs dispensed, extra blood and PBMCs collected, Ca/vitamin D intake check

   Week 1 Visit

   -Lab tests, AE, concomitant medications, Ca/vitamin D intake check

   Week 4 (1 Mo) Visit -Vital signs, labs (blood, urine), AE, concomitant medications, pen teaching, supplements and study drugs dispensed, extra blood and PBMCs collected, Ca/vitamin D intake check

   Week 8 (2 Mo) Visit

   -Vital signs, labs (blood, urine), AE, concomitant medications, pen teaching, supplements and study drugs dispensed, extra blood and PBMCs collected, Ca/vitamin D intake check

   Week 12 (3 Mo) Visit

   -Vital signs, labs (blood, urine), AE, concomitant medications, pen teaching, supplements and study drugs dispensed, extra blood and PBMCs collected, Ca/vitamin D intake check

   Week 20 (5 Mo) Visit -Vital signs, labs (blood), AE, concomitant medications, pen teaching, supplements and study drugs dispensed, extra blood collected, Ca/vitamin D intake check

   Week 24 (6 Mo) Visit

   -Vital signs, labs (blood, urine), AE, concomitant medications, pen teaching, supplements and study drugs dispensed, extra blood and PBMCs collected, Ca/vitamin D intake check

   Week 36 (9 Mo) Visit

   -Vital signs, labs (blood, urine), AE, concomitant medications, pen teaching, supplements and study drugs dispensed, extra blood and PBMCs collected, Ca/vitamin D intake check

   Week 48 (11 Mo) Visit

   -DXA, TBS, history, physical exam, vital signs, labs (blood, urine), AE, concomitant medications, extra blood and PBMCs collected, Ca/vitamin D intake check

5.Study Analysis

Statistical Analysis Plan

Statistics will include descriptive as well as analytic approaches. The intention-to-treat (ITT) approach will be used, with all randomized men included in the analysis. Complete follow-up data will be collected on every randomized subject, regardless of adherence. 2o per-protocol analyses will be done, limited to those who remained on medication and those with complete data. All statistical testing will be performed at nominal 0.05 level without adjustments for multiple comparisons.

Analysis of Primary Endpoint

To determine the effects of 11 months of treatment with TPTD+cinacalcet compared to TPTD+PBO on LS BMD (primary endpoint) Testing the 1o hypothesis for the effect of the 2 treatment arms on the % change in LS BMD will use a t-test with a two-sided significance level of 0.05. The extent of missing data will be reported in all statistical analyses. Overall missing data rates are expected to be low since the investigators will make every attempt to obtain BMDs at 11 months for all men, regardless of medication use. 1o analyses will be unadjusted. Using standard statistical methods and means and SDs from published TPTD studies, the effect size (true difference in means between treatment groups) that can be detected based on a t-test comparison between treatment groups of the change in LS BMD with a fixed sample size of 24/group was calculated. Even if 20% of the subjects were lost to follow-up and did not contribute 11-month LS BMD data, with a sample size of 40 the study is powered to detect a between-group difference as small as 4.0%. A difference between treatment regimens of ~4% (e.g., mean LS BMD increase in TPTD+PBO of 5% vs 9% increase in the combination group) would be an effect size for BMD in the range that would be clinically promising and support pursuing further studies of this combination therapy for osteoporosis.

Analysis of Secondary Endpoints

To determine the effects of 11 months of treatment with TPTD+cinacalcet compared to TPTD+PBO on FN BMD and levels of the bone formation marker P1NP (secondary endpoints).

A similar approach will be taken for FN BMD and for the logarithm of the P1NP change as will be taken for the primary endpoint above. On an exploratory basis, changes in TBS from baseline to study end will be analyzed as BMD is. All hypotheses will be tested at the nominal 0.05 2-sided significance level, with no formal adjustment for multiple comparisons. In the analysis of 2o outcomes and in other 2o analyses, it is recognized that this might increase type 1 error rates, due to multiple testing. To alleviate that concern, 1o and 2o endpoints will be clearly distinguished, as well as exploratory analyses. Consistency among multiple endpoints will be looked and caution will be exercise in interpreting marginally significant findings, particularly unexpected results not motivated by a priori hypotheses. The extent of missing data will be reported in all statistical analyses. Overall missing data rates are expected to be low since every attempt will be made to obtain BMDs at 11 months and P1NP at 3 months for all men, regardless of medication use. 1o analyses will be unadjusted.

This study has 80% power (with an alpha=0.05) to detect a between-group difference in change in FN BMD as small as 3.5%. Since effects of TPTD on FN BMD in short-term studies are small, it is recognized that +3.5% may be an ambitious difference between treatments for hip BMD. However, the point estimates may give an indication of whether the combination has superior effects on BMD at the hip and help investigators to plan future studies of this combination.

The distribution of P1NP change is non-Gaussian in multiple studies, requiring log transformation (log ratio) and back-transformation for presentation. Using data from the PaTH (Parathyroid Hormone and Alendronate for Osteoporosis ) trial of the 3-month change in P1NP, the back-transformed mean change (95% CI) was +148% (117%, 183%). Based on the SD of the log ratio in PaTH, a sample size of 40 (20/group, assuming 20% non-completers) will provide 80% power with alpha=0.05 to detect a difference of +137% (e.g., an increase from 148% to 285%) between P1NP responses of men treated with TPTD+cinacalcet vs TPTD+PBO.

ELIGIBILITY:
Inclusion Criteria:

* DXA BMD T-score < or = -2.0 at either lumbar spine (LS), femoral neck (FN) or total hip (TH) sites; or DXA BMD T-score < or = -1.5 with at least one additional important clinical risk factor for osteoporotic fracture [e.g., fragility fracture after age 50 years; parental history of hip fracture; history of hypogonadism, prior glucocorticoid therapy (>3 months prior), current smoking, prevalent vertebral fracture(s), or prior hyperthyroidism on stable treatment]
* At least 2 LS vertebral levels with reliable BMD values (i.e., at least 2 without compression or hardware)

Exclusion Criteria:

* Metabolic bone disease other than osteoporosis (e.g., Paget's disease, hyperparathyroidism)
* Any osteoporosis drug therapy within 12 months; any prior course of TPTD for > or = 3 months; any history of IV bisphosphonate therapy; oral bisphosphonate therapy exceeding 3 months in past 2 years; oral bisphosphonate treatment exceeding 2 years ever; or use of denosumab (within the past 3 years or > 3 or = injections ever).
* Oral glucocorticoid use (> or = 5 mg prednisone) taken within 3 months prior to enrollment
* Hypercalcemia (albumin-corrected serum [Ca] >10.2 mg/dL), hypocalcemia (albumin-corrected serum [Ca] <8.8 mg/dL), elevated intact PTH level, or hypercalciuria (urinary Ca >300 mg/24 hours) at screening
* 25 OH vitamin D levels <20 ng/ml or >80 ng/ml at screening
* Estimated glomerular filtration rate < 30 ml/min (chronic kidney disease (CKD) stage 4 or 5)
* Cancer within past 5 years except for non-melanomatous skin cancers
* History of skeletal radiation, prior history of osteosarcoma or bone metastases
* Substance abuse (>3 drinks/day), liver disease or impaired liver function (abnormal liver function tests defined as greater than 3 times the upper limit of normal), known cirrhosis, malabsorption
* Poorly controlled diabetes (A1c >9.0%) or current thiazolidinedione therapy
* Drugs metabolized through CYP2D6 (e.g., flecainide, tricyclic antidepressants) and strong inducers or inhibitors of CYP3A4 (e.g., itraconazole, ketoconazole)
* Testosterone therapy with dose change within last 12 months; or androgen deprivation therapy within 12 months
* Thyrotropin (TSH) level < 0.01
* Congenital long QT syndrome, history of QT interval prolongation, family history of long QT syndrome or sudden cardiac death, and other conditions that predispose to QT interval prolongation and ventricular arrhythmia
* Hypersensitivity to teriparatide or any excipients in Forteo
* Use of other Ca-lowering drugs (e.g., calcitonin, bisphosphonates, denosumab)
* Moderate to severe hepatic impairment
* High risk for active urolithiasis, defined as having passed a kidney stone clinically within the last 5 years
* Upper gastrointestinal (GI) bleeding with a history of a clinical episode of upper GI bleeding within last 10 years that was note definitively treated by a surgical procedure
* Orthostatic hypotension or a known history of orthostatic hypotension documented in the chart or provided by the patient upon clinical history-taking
* Impaired cardiac function either diagnosed symptomatic heart failure requiring medical therapy

Ages: 60 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Effects of treatment with TPTD+cinacalcet compared to TPTD+PBO on lumbar spine BMD in men with low bone mass | 48 weeks
  Hypothesis 1a proposes that BMD responses to combined TPTD+cinacalcet are greater than those induced by TPTD+PBO. LS BMD typically responds quickly and robustly to TPTD and is the 1o endpoint of the trial. DXA measurements will be performed and analyzed by standard protocols at baseline and at the end of the trial. Subjects will be treated for 11 months (48 weeks). All subjects will receive Ca and vitamin D3 supplements throughout the trial. The percentage change in LS BMD from baseline to 48 week/11 months of treatment will be the variable/endpoint that is calculated.

SECONDARY OUTCOMES:
Effects of treatment with TPTD+cinacalcet compared to TPTD+PBO on serum P1NP in men with low bone mass | 48 weeks
  Hypothesis 1b proposes that serum P1NP (N-terminal pro-peptide of type 1 collagen), a highly sensitive marker of bone turnover and specifically of bone formation, will increase to a greater extent in men treated with TPTD+cinacalcet vs TPTD+PBO. Serum P1NP is the best validated biomarker of TPTD action and responds rapidly and robustly to anabolic therapy. This secondary endpoint will be assessed at the 3 month/12 week visit in the fasting state on morning lab tests (prior to study drug administration). The endpoint is a blood test of bone formation marker comparing results from Day 1/Randomization Visit to Study Visit at 3 months/12 weeks. The percentage change in this bone formation marker will be the variable that will constitute this secondary endpoint.
Effects of treatment with TPTD+cinacalcet compared to TPTD+PBO on femoral neck BMD in men with low bone mass | 48 weeks
  Hypothesis 1a also proposes femoral neck BMD responses to combined TPTD+cinacalcet are greater than those induced by TPTD+PBO. FN BMD responses tend to be smaller than LS BMD responses to TPTD and this aim will test whether the combination therapy (CaSR activation + PTH-R activation) will produce larger BMD responses at the FN site in men with low BMD. The percentage change in FN BMD from baseline to 48 week/11 months of treatment will be the variable/endpoint that is calculated.

OTHER OUTCOMES:
Pharmacodynamic responses to TPTD+cinacalcet and to TPTD+PBO in men with low bone mass | 48 weeks
  This outcome has two components testing 2 hypotheses. Hypothesis 2a proposes that serum Ca levels do not decrease to >5% below lower limits of normal in response to study drugs. Hypothesis 2b proposes that urinary Ca excretion does not exceed 350 mg/24 hrs in men treated chronically with study drugs. Hypothesis 2a will be in 2 ways: (1) PD testing done at Randomization Visit where serial blood samples (for serum Ca, PTH, phosphate, albumin) will be done at time 0, 2, 4, and 8 hrs after study drugs are given (acute PD). (2) Throughout the study PD responses will be assessed by measuring serum Ca levels (and albumin, phosphate, PTH) at every visit. This will assess chronic changes in serum minerals and PTH with 48 week/11 month treatment (chronic PD). 24 hr urine Ca is assessed at baseline and at defined times in full trial (chronic PD). Urine Ca is expected not to exceed 350 mg during the study. Each time-point of assessment will be compared to baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Dolores M. Shoback, MD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) sets will be shared. All IPD collected during the trial after de-identification will be shared. The types of Supporting Information that will be shared (in addition to IDP and Data Dictionaries) include Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report, and Analytic Code. The data will be available 6 months after the publication of the study, with no end date, and will be available to anyone who wishes to access the data and provides a methodologically sound proposal. The types of analyses that are planned in that proposal will be reviewed by the research study team of investigators, consultants and collaborators. To gain access to the data, requesting investigators will need to sign a Data Use Agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six (6) months after the trial data are published and then indefinitely afterwards
Access Criteria: All IDP data after deidentification collected during the trial will become available 6 months after the trial publication is published. This is a 5-year project commencing approximately July 1, 2019, and will continue through June 30, 2024, until all subject level data is collected and the trial interventions completed. Once study data are fully analyzed and published, then 6 months later, the IPD data sets and IPD Supporting Information will be available to other investigators.

DOCUMENTS (1):
  • Informed Consent Form (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT03994172/ICF_000.pdf